CLINICAL TRIAL: NCT04126668
Title: A Pharmacokinetic Study in Chinese Healthy Male and Female Volunteers to Investigate the Effect of Food on the Pharmacokinetics of CM082 Tablet.
Brief Title: A Study to Investigate the Food Effect on the Pharmacokinetics of CM082 Tablet in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AnewPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CM082-CA-I-106
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Advanced Malignant Solid Tumors
MeSH Terms: interventions — vorolanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1: fasted control → Period 2: fed control (Experimental): Period 1: administration of CM082 200 mg at 7:30am, without the breakfast；Period 2: administration of CM082 200 mg at 7:30am, 30 minutes after the breakfast
  Interventions: Drug: CM082 with fed or fasting
- Period 1: fed control → Period 2: fasted control (Experimental): Period 1: administration of CM082 200 mg at 7:30am, 30 minutes after the breakfast；Period 2: administration of CM082 200 mg at 7:30am, without the breakfast
  Interventions: Drug: CM082 with fed or fasting

INTERVENTIONS:
Drug: CM082 with fed or fasting — The two groups of subjects were given an equal dose of CM082 tablet (200 mg) after a single cross-over fasting or high-fat high-calorie diet in two different test cycles to examine the effect of food on the pharmacokinetics of CM082.

SUMMARY:
The main objective of this study is to evaluate the Effect of Food on the Pharmacokinetics of CM082 tablet.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the Effect of Food on the Pharmacokinetics of CM082 tablet in Chinese Healthy Volunteers. In addition, the safety of CM082 tablet in Chinese Healthy Volunteers who with High-fat meal or fasting state will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years;
* sex: male and female;
* body weight: Male ≥ 50 kg,female ≥ 45 kg, body mass index BMI (weight (kg)/height 2 (m2)) between 19-26 kg/m2 (including border);
* Healthy as judged by the investigator/subinvestigator based on the results of physical examinations and all lab tests;
* Abstinence or physical contraception approved by researchers must be approved during and within three months after the trial is completed; and no sperm and egg donation plan is available；
* Written informed consent;

Exclusion Criteria:

* Received any investigational drugs within 14 days before the screening test;
* Donated 200 mL of whole blood within 30 days before the screening test,or donated 200 mL of whole blood during the study or within 30 days after completion of the study;
* Females who are lactating, pregnant, potentially child-bearing, or willing to get pregnant during the study period;
* History of drug or food allergies;
* Abnormal blood pressure or pulse，Abnormal laboratory tests;
* Participated in other clinical trials within 3 months before screening;
* Smoking and drinking within 3 months before screening or test results of smoke, alcohol, and drug abuse are positive;
* Positive for HBsAg, Hepatitis C virus (HCV) antibody, HIV antibody or syphilis antibody;
* Clinically apparent disease/infection within 1 month before screening;
* The researchers determined that there were other conditions that were not suitable for the trial;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of CM082 | pre-dose(30minute),30min、1、1.5、2、2.5、3、3.5、4、4.5、5、6、8、10、12、24、36、48、72hour (after administration)
  The effect of food on Cmax after high fat diet and fasting Blood sampling over a 72 hour period post dose in all dosing sessions
Area under the plasma concentration versus time curve (AUC) of CM082 | pre-dose(30minute),30min、1、1.5、2、2.5、3、3.5、4、4.5、5、6、8、10、12、24、36、48、72hour (after administration)
  The effect of food on AUC after high fat diet and fasting Blood sampling over a 72 hour period post dose in all dosing sessions
Time of maximum concentration（Tmax）of CM082 | pre-dose(30minute),30min、1、1.5、2、2.5、3、3.5、4、4.5、5、6、8、10、12、24、36、48、72hour (after administration)
  The effect of food on Tmax after high fat diet and fasting Blood sampling over a 72 hour period post dose in all dosing sessions
Half life（T1/2）of CM082 | pre-dose(30minute),30min、1、1.5、2、2.5、3、3.5、4、4.5、5、6、8、10、12、24、36、48、72hour (after administration)
  The effect of food on T1/2 after high fat diet and fasting Blood sampling over a 72 hour period post dose in all dosing sessions

SECONDARY OUTCOMES:
Percentage of adverse events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 months
  Percentage of adverse events as assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: zourong ruan, Study Chair — the Second Affiliated Hospital of Zhejiang University Medical College
Locations (1):
- The 1st Phase Clinical Research Center of the Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No